CLINICAL TRIAL: NCT03798093
Title: Hemodynamic Changes With Umbilical Cord Milking in Nonvigorous Newborns
Brief Title: Echocardiography Sub-Study of the Umbilical Cord Milking in Non-Vigorous Infants Trial (MINVI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director, Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: MINVI Echo Study
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Birth Asphyxia
Keywords: Umbilical Cord Milking; Immediate Cord Clamping; Resuscitation
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Crossover
Who Masked: Outcomes Assessor
Masking Description: Cardiac research sonographers that obtained study measurements were blinded to the study intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): The delivering practitioner will place the newborn below the level of the incision (at the edge of the table) at C/S and a second team member will milk the cord four times. For vaginal delivery, the delivering obstetrician, midwife or perinatal provider will hold the infant against their body or place the infant on the mother's abdomen and the cord will be milked either four times by the obstetrical provider or by a second team member. For the cord milking procedure, the obstetrical provider will milk the entire length of umbilical cord over two seconds, repeating three additional times as described previously. This time is not significantly different from the time for Early Cord Clamping as we have demonstrated in our previous trials.
  Interventions: Procedure: Umbilical Cord Milking
- Early Cord Clamping (Active Comparator): This will occur by clamping the umbilical cord as soon as possible. Since both Early Cord Clamping and Umbilical Cord Milking will occur after a brief assessment, it is important to note that the cord clamping time will be longer than in previously conducted preterm trials (average 20 seconds) which performed the intervention on all subjects regardless of whether or not they were vigorous. In all cases, the cord clamping time will be documented to ensure consistency.
  Interventions: Procedure: Early Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 15-20 seconds.
  Arms: Umbilical Cord Milking
Procedure: Early Cord Clamping — The umbilical cord is clamped within 60 seconds of delivery.
  Arms: Early Cord Clamping

SUMMARY:
Non-vigorous infants enrolled in the MINVI trial will be approached for consent for ongoing data collection. As part of the data collection, an optional echocardiogram will be performed if the parent consents.

DETAILED DESCRIPTION:
Non-vigorous infants enrolled in the MINVI trial will be approached for consent for ongoing data collection. As part of the data collection, an optional echocardiogram will be performed if the parent consents. The consent will have a check box to indicate if they consent to the additional test.

Echocardiographic measurements will be performed on all infants at 12 hours +/- 6 hours of age by our research sonographers who are blinded to infant randomization. Measurements will be taken according to a standard operating procedure to assess systemic blood flow, by superior vena cava (SVC) flow (ml/kg/min), right ventricular output (ml/kg/min), left ventricular output (LVO) (ml/kg/min), measures of left and right ventricular tissue Doppler and strain imaging. These measurements will be performed offline at a later time. Data will be entered into REDCap.

If any structural abnormalities are found, the attending pediatrician will be notified of the abnormal echocardiogram. The consent will clearly state that this echo is not for diagnostic purposes. Any additional studies including an official complete echocardiogram and or cardiology consultation will be left to the discretion of the attending pediatrician, as he/she deems necessary

ELIGIBILITY:
Inclusion Criteria:

• Non-vigorous newborns born between 35-42 weeks gestation.

Exclusion Criteria:

* Known major congenital or chromosomal anomalies of newborn.
* Known cardiac defects other than small atrial septal defect (ASD), ventricular septal defect (VSD) and patent ductus arteriosus (PDA).
* Complete placental abruption/cutting through the placenta at time of delivery.
* Monochorionic multiples
* Cord anomaly (i.e. cord avulsion or true knot)
* Presence of non-reducible nuchal cord
* Perinatal providers unaware of the protocol
* Incomplete delivery data
* Infants born in extremis, for whom additional treatment will not be offered.

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katheria A, Mercer J, Poeltler D, Morales A, Torres N, Lakshminrusimha S, Singh Y. Hemodynamic Changes with Umbilical Cord Milking in Nonvigorous Newborns: A Randomized Cluster Cross-over Trial. J Pediatr. 2023 Jun;257:113383. doi: 10.1016/j.jpeds.2023.03.001. Epub 2023 Mar 11. PMID 36914049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at two maternity hospitals involved in a cluster crossover randomization trial of non-vigorous infants at birth randomized to perform umbilical cord milking in the initial period (January 2019-January 2020) and early cord clamping in the crossover period (February 2020- March 2021). Participants were enrolled in this study upon parental consent for a neonatal echocardiogram in the first 12 hours of life. Participants enrolled in periods 1 & 2 are unique participants.
Pre-assignment Details: The two hospitals who participated in the echocardiography sub-study and were both randomized to implement umbilical cord milking in the initial period (Period 1) and randomized to implement early cord clamping in the cross over period (Period 2).
Units Other Than Participants: Hospital
Groups:
- Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Neonate: In the first study period infants assessed as non-vigorous at delivery had the umbilical cord is grasped by the obstetric provider, and blood was pushed toward the infant 4 times before the cord is clamped.
  In the second study period infants assessed as non-vigorous at delivery had the umbilical cord clamped by 60 seconds of life.
- Early Cord Clamping Then Umbilical Cord Milking - Neonate: In the first study period infants assessed as non-vigorous at delivery had the umbilical cord clamped as soon as possible and within 60 seconds of delivery. In the second study period umbilical cord was grasped by the obstetric provider, and blood was pushed toward the infant 4 times before the cord is clamped.
Period: Initial Randomized Intervention
Arm/Group | Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Neonate | Early Cord Clamping Then Umbilical Cord Milking - Neonate
Started | 106; 2 Hospital | 0; 0 Hospital (None of the hospital sites randomized to perform early cord clamping then umbilical cord milking recruited participants for this substudy.)
Completed | 106; 2 Hospital | 0; 0 Hospital
Not Completed | 0; 0 Hospital | 0; 0 Hospital
Period: Crossover Randomized Intervention
Arm/Group | Umbilical Cord Milking Then Early Cord Clamping Site Randomization - Neonate | Early Cord Clamping Then Umbilical Cord Milking - Neonate
Started | 121; 2 Hospital (In this study design the participants recruited in the initial study period with treatment of umbilical cord milking did not continue on to the crossover period. In the cross over period hospital sites recruited new participants with a target enrollment equivalent to the site's recruitment in the initial study period and performed early cord clamping in the second study period.) | 0; 0 Hospital (None of the hospital sites randomized to perform early cord clamping then umbilical cord milking recruited participants for this substudy.)
Completed | 121; 2 Hospital | 0; 0 Hospital
Not Completed | 0; 0 Hospital | 0; 0 Hospital

BASELINE CHARACTERISTICS:
Groups:
- Umbilical Cord Milking - Neonate: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. Both participating hospitals were randomized to perform umbilical cord milking as the first intervention in the primary trial. Maternal data is presented for all participating mothers. Only unique participants are presented.
- Early Cord Clamping - Neonate: The umbilical cord is clamped as early as possible and within 60 seconds of delivery. Both participating hospitals were randomized to perform early cord clamping as the second intervention in the primary trial. Maternal data is presented for all participating mothers. Only unique participants are presented.
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate | Total
Number analyzed (Participants) | 106 | 121 | 227
Age, Continuous [Median (Inter-Quartile Range); unit: weeks]
  Neonatal Birth Gestational Age | 40 [39 to 40] | 39 [38 to 40] | 39 [38 to 40]
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Maternal Age | 31 [27 to 33] | 30 [25 to 36] | 31 [27 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Neonatal Sex: Female | 45 | 50 | 95
  Neonatal Sex: Male | 61 | 71 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Neonatal Ethnicity: Hispanic or Latino | 45 | 52 | 97
  Neonatal Ethnicity: Not Hispanic or Latino | 60 | 69 | 129
  Neonatal Ethnicity: Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Maternal Ethnicity: Hispanic or Latino | 39 | 44 | 83
  Maternal Ethnicity: Not Hispanic or Latino | 66 | 77 | 143
  Maternal Ethnicity: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Neonatal Race: American Indian or Alaska Native | 0 | 0 | 0
  Neonatal Race: Asian | 5 | 7 | 12
  Neonatal Race: Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Neonatal Race: Black or African American | 1 | 6 | 7
  Neonatal Race: White | 52 | 50 | 102
  Neonatal Race: More than one race | 28 | 34 | 62
  Neonatal Race: Unknown or Not Reported | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Maternal Race: American Indian or Alaska Native | 1 | 0 | 1
  Maternal Race: Asian | 5 | 11 | 16
  Maternal Race: Native Hawaiian or Other Pacific Islander | 0 | 4 | 4
  Maternal Race: Black or African American | 2 | 8 | 10
  Maternal Race: White | 64 | 58 | 122
  Maternal Race: More than one race | 13 | 16 | 29
  Maternal Race: Unknown or Not Reported | 21 | 24 | 45
Maternal Diabetes [Count of Participants; unit: Participants] — Number of neonates delivered by a mother with diabetes during pregnancy.
  Participants | 14 | 16 | 30
Maternal Hypertension or Pre-eclampsia [Count of Participants; unit: Participants] — Number of neonates delivered by a mother who experienced hypertension or pre-eclampsia during pregnancy.
  Participants | 14 | 17 | 31
Maternal Intrauterine Inflammation/Infection [Count of Participants; unit: Participants] — Number of neonates delivered by a mother diagnosed with intrauterine inflammation or intrauterine infection.
  Participants | 19 | 27 | 46
Maternal Group B Streptococcus Positive [Count of Participants; unit: Participants] — Number on infants born to a mother with positive group B streptococcus culture prior to delivery
  Participants | 19 | 18 | 37
Maternal General Anesthesia [Count of Participants; unit: Participants] — Number of neonates delivered by a mother who was administered general anesthesia at the time of delivery.
  Participants | 2 | 7 | 9
Multiple Gestation [Count of Participants; unit: Participants] — Number of neonates delivered by a mother with a multiple gestation pregnancy
  Participants | 1 | 3 | 4
Delivery of the Neonate via Cesarean Section [Count of Participants; unit: Participants] | 49 | 53 | 102
Number of hours Membranes were Ruptured Before Delivery [Median (Inter-Quartile Range); unit: hours] | 7 [2 to 17] | 6 [0 to 14] | 6 [1 to 14]
Neonatal Weight at Birth [Mean (Standard Deviation); unit: grams] | 3443 (543) | 3386 (584) | 3413 (564)
Neonates with Poor Color at Birth [Count of Participants; unit: Participants] — In the first 15 seconds of life the infant's skin color was assessed by the obstetric provider and assessment of poor color (pale, dusky, cyanotic) was reported on the study specific case report form.
  Participants | 105 | 118 | 223
Neonates with Poor Tone at Birth [Count of Participants; unit: Participants] — In the first 15 seconds of life the infant's tone was assessed by the obstetric provider and assessment of poor infant tone was reported on the study specific case report form.
  Participants | 104 | 117 | 221
Neonates with Poor Respiratory Effort at Birth [Count of Participants; unit: Participants] — In the first 15 seconds of life the infant is assessed for respiratory effort by the obstetric provider and assessment of poor respiratory effort it reported on the study specific case report form.
  Participants | 103 | 120 | 223
Neonates Treated with Therapeutic Hypothermia [Count of Participants; unit: Participants] — Number of neonates treated with therapeutic hypothermia (cooling to 33.5 degrees Celsius) for 72 hours and initiated in the first 6 hours of life.
  Participants | 5 | 17 | 22
Neonates Treated with Cardiac Inotropes [Count of Participants; unit: Participants] | 3 | 5 | 8
Neonates Treated with Volume Expanders [Count of Participants; unit: Participants] | 20 | 30 | 50
Time of Echocardiogram Exam from Neonate's Time of Birth [Median (Inter-Quartile Range); unit: hours] | 13 [10 to 17] | 15 [11 to 17] | 15 [11 to 17]
Venous Cord Blood Gas pH [Mean (Standard Deviation); unit: no units] — Population: Venous cord gas values reported for all neonates with results available for venous cord blood pH results.
  no units
    number analyzed (Participants) | 84 | 96 | 180
    (all) | 7.266 (.095) | 7.234 (.122) | 7.249 (.111)
Venous Cord Blood Gas Base Excess [Mean (Standard Deviation); unit: mEq/L] — Population: Venous cord gas values reported for all neonates with results available for venous cord blood base excess results.
  mEq/L
    number analyzed (Participants) | 84 | 96 | 180
    (all) | -6.60 (3.12) | -7.31 (4.22) | -6.98 (3.75)
Arterial Cord Blood Gas pH [Mean (Standard Deviation); unit: no units] — Population: Arterial cord gas values reported for all neonates with results available arterial cord blood pH results.
  no units
    number analyzed (Participants) | 70 | 80 | 150
    (all) | 7.173 (.104) | 7.125 (.140) | 7.148 (.127)
Arterial Cord Blood Gas Base Excess [Mean (Standard Deviation); unit: mEq/L] — Population: Venous cord gas values reported for all neonates with results available for arterial cord blood base excess results.
  mEq/L
    number analyzed (Participants) | 70 | 80 | 150
    (all) | -8.74 (3.96) | -9.77 (5.11) | -9.29 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Output
Description: Left ventricular output measurements taken by cardiac ultrasound.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Umbilical Cord Milking - Neonate: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. Both participating hospitals were randomized to perform umbilical cord milking as the first intervention in the primary trial.
- Early Cord Clamping - Neonate: The umbilical cord is clamped as early as possible and within 60 seconds of delivery. Both participating hospitals were randomized to perform early cord clamping as the second intervention in the primary trial.
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
mL/kg/min | 225 (64) | 187 (52)
Statistical Analysis 1: Comparison: Umbilical Cord Milking - Neonate vs Early Cord Clamping - Neonate; Test type: Superiority; p = 0.08, Regression, Linear; least squares = -0.112, 95% CI 2-sided [-29.3 to 1.7]

2. Secondary Outcome: Neonatal Right Ventricular Output
Description: Obtained from the modified short axis view of the neonatal echocardiogram performed at 12 hours of life ± 6 hours.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Umbilical Cord Milking - Neonate: At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped.
- Early Cord Clamping - Neonate: The umbilical cord is clamped as early as possible and within 60 seconds of delivery.
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
mL/kg/min | 284 (88) | 222 (95)

3. Secondary Outcome: Neonatal Superior Vena Cava Flow
Description: superior vena cava (SVC) flow (Diameter obtained from the infraclavicular view (hybrid view) and doppler assessment from the subcostal view of the neonatal echocardiogram exam performed at 12 hours of life ± 6 hours.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
mL/kg/min | 100 (36) | 86 (40)

4. Secondary Outcome: Neonatal Peak Systolic Strain
Description: This measurement reflects the deformation (strain) of the heart muscle during systole (the phase of the heartbeat when the heart contracts) relative to its original length. More negative values indicate better myocardial function while values closer to 0 suggest impaired myocardial function.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
percent | -17 (3) | -22 (3)

5. Secondary Outcome: Neonatal Peak Systolic Velocity
Description: Measure of left and right ventricular peak systolic tissue doppler velocity on neonatal echocardiogram performed at 12 hours of life ± 6 hours.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
meters/second | .06 (.02) | .07 (.02)

6. Other Pre Specified Outcome: Tricuspid Annular Plane Systolic Excursion Measurement in Neonate
Description: Assessment of tricuspid annular plane systolic excursion in the neonate by echocardiogram performed at 12 hours of life ± 6 hours
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
mm | 9.04 (2.2) | 9.65 (1.7)

7. Other Pre Specified Outcome: Number of Neonates With a Patent Ductus Arteriosus
Description: Diagnosis of patent ductus arteriosus in neonate by echocardiogram with diameter measurement and direction of flow.
Time Frame: 12 ± 6 hours of life
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
Participants | 88 | 110

8. Other Pre Specified Outcome: Neonatal Direction of Ductal Shunt
Description: Direction of ductal shunt in neonate assessed by echocardiogram which was performed at 12 hours of life ± 6 hours.
Time Frame: 12 ± 6 hours of life
Population: Direction of shunt assessed only for neonates with a patent ductus arteriosus present.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 87 | 108
Participants
  All left to right | 59 | 80
  All right to left | 0 | 1
  Bidirectional | 28 | 27

9. Post Hoc Outcome: Diameter of Neonatal Ductus Arteriosus
Description: Diameter of neonatal ductus arteriosus assessed by echocardiogram which was performed at 12 hours of life ± 6 hours
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
cm | 0.19 (0.10) | 0.20 (0.10)

10. Post Hoc Outcome: Neonatal Peak Pulmonary Artery Pressure
Description: Neonatal peak pulmonary artery pressure as measured by echocardiogram at 12 hours of life ± 6 hours.
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
mm Hg | 27 (15) | 27 (14)

11. Post Hoc Outcome: Mean Neonatal Blood Pressure at Time of Echocardiogram
Description: blood pressure measurement obtained at the time of cardiac ultrasound examination
Time Frame: 12 ± 6 hours of life
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
g/dL | 45 (7) | 46 (7)

12. Post Hoc Outcome: Median Neonatal Hemoglobin
Description: Single neonatal hemoglobin measurement obtained between 12 and 48 hours of life either as part of standard care or obtained with parental written consent
Time Frame: 12 to 48 hours of life
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
Number analyzed (Participants) | 106 | 121
g/dL | 17.6 (2.1) | 16.5 (2.4)

ADVERSE EVENTS:
Time Frame: Assessed from neonate's birth to discharge home up to 180 days of life
Description: Adverse events were assessed for all neonate participants enrolled in the study and were collected from delivery to discharge home or up to 180 days of life.
  All known adverse events are reported in the All-Cause Mortality, serious adverse events, and other adverse events tables.
Arm/Group | Umbilical Cord Milking - Neonate | Early Cord Clamping - Neonate
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/121
Other Adverse Events (participants affected / at risk) | 0/106 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03798093/Prot_SAP_000.pdf